CLINICAL TRIAL: NCT02225366
Title: Induction of Antitumor Response in Melanoma Patients Using the Antimicrobial Peptide LL37
Brief Title: Intratumoral Injections of LL37 for Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0422; 5P50CA093459-08 (NIH); NCI-2014-02012 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic; Antimicrobial peptide; LL37; Photographs
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intra-Tumoral Injection of LL37 (Experimental): LL37 administered intratumorally in cutaneous or subcutaneous tumors at least 1 cm in diameter. Patients will receive weekly intratumoral injections of LL37 for up to 8 weeks. The injections will be given every 7 days (+/- 48 hours). Starting dose 250 µg/tumor.
  Interventions: Biological: LL37; Other: Photographs

INTERVENTIONS:
Biological: LL37 — Starting dose 250 µg/tumor. The injections will be given every 7 days for up to 8 weeks.
Other: Photographs — Tumors measured and photographed one week before receiving LL37, and again at 4 weeks after LL37. Then photographs of the LL37 injected sites taken at 8 weeks.

SUMMARY:
The goal of this clinical research study is to find the appropriate dose of LL37 that can be given to patients with melanoma. Researchers also want to learn if LL37 can stimulate the immune system to help control the disease.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of LL37 based on when you join this study. Up to 4 dose levels of LL37 will be tested. Up to 2 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of LL37 is found.

Study Drug Administration:

One (1) time a week for 8 weeks, LL37 will be injected into 2-4 tumors. The injections will be done in the clinic.

Study Visits:

Within 1 week before your first study drug injection:

* You will have a physical exam.
* You will have a punch biopsy of a tumor. To collect a punch biopsy, the area of skin is numbed with anesthetic and a small cut is made to remove all or part of the affected tissue.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* The tumors will be measured and photographed. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are tumors on your face.

On Day 1:

* You will have a physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.

On Day 2, you will have a punch biopsy of one of the injected tumors.

At Weeks 1, 2, 3, 4, 5, 6, 7, and 8:

* You will have a physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* At Weeks 1, 3, and 5 and 7, blood (about 4 tablespoons) will be drawn to study your immune response to LL37.

At Week 4, you will have a punch biopsy of one of the injected tumors and one of the tumors that you did not have an injection in. Photos of the tumors will be taken to show if the disease has responded to the study drug.

At Week 8:

* Photos of the LL37 injected sites will be taken to show if the disease has responded to the study drug.
* You will have CT scans to check the status of the disease.

Length of Treatment:

You will receive up to 8 weeks of study treatment. You will be taken off study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Off-Study Visit:

If you have to stop the study treatment earlier than planned because the disease got worse or you had intolerable side effects:

* You will have a physical exam.
* The tumors will be photographed and measured.
* Blood (about 4 teaspoons) will be drawn for routine tests and to study your immune response to LL37.
* You will have CT scans to check the status of the disease.
* You will have a punch biopsy of one of the injected tumors.

These off-study procedures will be completed within 14 days after your last dose of study treatment. You will be contacted by phone or clinic visit at 30 days (+/- 7 days) after your last dose to follow up on any drug-related toxicities which were present at the end of study.

Follow-Up:

Within 2 weeks after your last study drug dose and every 8-12 weeks after that, you will have scans to check the status of the disease. Your doctor will decide what type of scans you will have.

After your last study drug dose, at your routine clinic visits every 3 months for 1 year, the study staff will ask you about the status of disease, if possible. If you do not plan to continue to receive medical care at MD Anderson, the study staff will contact you by phone, email, or letter to ask about the status of disease. The calls should last about 5 minutes.

This is an investigational study. LL37 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 36 participants will be treated in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented metastatic melanoma with at least 3 cutaneous lesions measuring over 5mm diameter. At least two lesions must be at least 10mm in diameter to serve as the injected disease. At least one other lesion measuring at least 5mm in diameter may serve as the non-injected lesion that will be measurable disease. Patients will have stage IIIB or IIIC (in-transit lesions with or without nodal metastases) or stage IV M1A disease with cutaneous or nodal lesions assessable for administration of LL37. Patients are only eligible if their melanoma deposits are not amenable to complete surgical excision. Skin lesions that are 5mm or greater are deemed measurable however lesions that are at least 10mm in diameter will be preferentially utilized for LL37 injection.
2. Age greater than or equal to 18 years
3. Clinical performance status of ECOG 0-2 within 30 days of signing informed consent.
4. Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
5. Platelet count greater than or equal to 100,000/mm^3
6. WBC >/=3000/mm^3
7. Serum ALT and AST less than three times the upper limit of normal
8. Serum creatinine </= 2.0 mg/dl
9. Seronegative for HIV antibody
10. Patients with a negative pregnancy test (urine or serum) must be documented within 28 days of starting treatment for women of childbearing potential (WOCBP).
11. Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, IUD, or sponge plus spermicide. Abstinence is an acceptable form of birth control.

Exclusion Criteria:

1. Active autoimmune disease requiring disease modifying therapy.
2. Concurrent systemic steroid therapy
3. Any form of active primary or secondary immunodeficiency
4. Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years.
5. History of immunization with LL37
6. Active systemic infections requiring intravenous antibiotics
7. Prior systemic therapy, radiation therapy, or surgery within 28 days of starting study treatment
8. Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N. Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: This cohort received starting dose of 250 ug/tumor injection once a week
- Cohort 2: This cohort received 500 ug/tumor injection once a week
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Optimal Biological Dose (OBD) of LL37 Based Upon Toxicity
Description: Dose Limiting Toxicity defined as: a. Any grade 3 or 4 non-hematologic toxicity regardless of duration, except: Grade 3 skin reactions at injection sites - Grade 3 fever b. Grade 4 thrombocytopenia c. Grade 4 neutropenia lasting >2 weeks or associated with infection.
Time Frame: once a week, up to 8 weeks duration
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

2. Secondary Outcome: Number of Participants With Antitumor Immune Response of Intra-Tumoral Injection of LL37
Description: Response defined as experiencing either an immune-related complete or partial response (irCR or irPR), and the association between response and disease characteristics and T-cell responses will be assessed using logistic regression.
Time Frame: Radiologic evaluations in the form of CT scans of affected disease sites will be performed every 8 weeks (+/- 14 days) while on study, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: adverse events were collected every week at the time of the injections for up to 8 weeks, All-Cause Mortality was assessed up to 14 months
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=1)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Lymphocyte Count Decrease (Blood and lymphatic system disorders) | 0 | 1
White blood cell decrease (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increase (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT02225366/Prot_SAP_000.pdf